CLINICAL TRIAL: NCT06049433
Title: Prevention of Perinatal Depression Among At-risk Individuals Through Integration of a Multimedia, Web-based Intervention Within the Healthcare System
Brief Title: Maternal Mental Health Access - MaMa
Acronym: MaMa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Gwen Latendresse, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 00159109; RF1NR020841 (NIH)
Record Dates: First submitted 2023-08-23; First posted 2023-09-22 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Postpartum Depression; Perinatal Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Abortion, Legal; DMAC2L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Choice 1 (Other): Options; On-Demand (OD) alone or On-Demand (OD) with a facilitated discussion board (DB)
  Interventions: Behavioral: Maternal Mental Health Access for Postpartum Depression- Prevention and UPLIFT- intervention; Behavioral: On-Demand + Discussion board (DB)
- Choice 2 (Other): Options:
  On-Demand (OD) + Discussion board (DB) or OD + Video Conference (VC)
  Interventions: Behavioral: Maternal Mental Health Access for Postpartum Depression- Prevention and UPLIFT- intervention; Behavioral: Arm 2; Behavioral: On Demand (OD) + Video Conference (VC)
- Choice 3 (Other): Options; Om-Demand (OD) or On-Demand (OD) + Video Conference (VC)
  Interventions: Behavioral: Maternal Mental Health Access for Postpartum Depression- Prevention and UPLIFT- intervention; Behavioral: Arm 3; Behavioral: On Demand (OD) + Video Conference (VC)

INTERVENTIONS:
Behavioral: Maternal Mental Health Access for Postpartum Depression- Prevention and UPLIFT- intervention — The intervention uses a standardized, manualized program (UPLIFT - Using Practice and Learning to Increase Favorable Thoughts) based on Mindfulness-Based Cognitive Behavioral Therapy (MBCT) in the prevention of depression in various populations and settings. MBCT can be delivered individually and in groups and via electronic platforms, in diverse populations. We have adapted UPLIFT for this study, based on input from focus groups and in response to the ongoing pandemic, and under the direction of our team's mental health professionals. Adaptations include access to asynchronous, on-demand multi-media MBCT content (digital audio-video files and downloadable content),
  Other Names: Arm 1; On-Demand (OD)
Behavioral: On-Demand + Discussion board (DB) — Adaptations include access to asynchronous, on-demand multi-media MBCT content (digital audio-video files and downloadable content), as well as synchronous Videoconference (VC) reduced from 8 weekly one-hour sessions to 4 one-hour sessions every two weeks. a discussion board with the potential to build a sense of community in a similar way that synchronous VC groups provide.
  Arms: Choice 1
Behavioral: Arm 2 — The intervention uses a standardized, manualized program (UPLIFT - Using Practice and Learning to Increase Favorable Thoughts) based on Mindfulness-Based Cognitive Behavioral Therapy (MBCT) in the prevention of depression in various populations and settings. MBCT can be delivered individually and in groups and via electronic platforms, in diverse populations. On-demand multi-media MBCT content (digital audio-video files and downloadable content)
  Other Names: On-Demand (OD) + Discussion Board (DB)
  Arms: Choice 2
Behavioral: On Demand (OD) + Video Conference (VC) — on-demand multi-media MBCT content (digital audio-video files and downloadable content), as well as synchronous Videoconference (VC) reduced from 8 weekly one-hour sessions to 4 one-hour sessions every two weeks. A discussion board with the potential to build a sense of community in a similar way that synchronous VC groups provide.
  Arms: Choice 2
Behavioral: Arm 3 — The intervention uses a standardized, manualized program (UPLIFT - Using Practice and Learning to Increase Favorable Thoughts) based on Mindfulness-Based Cognitive Behavioral Therapy (MBCT) in the prevention of depression in various populations and settings.
  Other Names: On Demand (OD)
  Arms: Choice 3
Behavioral: On Demand (OD) + Video Conference (VC) — Access to asynchronous, on-demand multi-media MBCT content (digital audio-video files and downloadable content), as well as synchronous Videoconference (VC)
  Arms: Choice 3

SUMMARY:
This hybrid effectiveness-implementation project will allow the team to evaluate and refine implementation in preparation for future multisite trials to ultimately move the Evidence-Based Intervention (EBI) to scale among diverse populations. The plan is to enroll 120 at-risk pregnant and postpartum women from rural, urban, and Latino populations. Using a randomized preference design to also evaluate patient and sociocultural factors in participation and symptom trajectory.

Using the Implementation Research Logic Model, the team will evaluate the implementation feasibility and acceptability of a remote-access and on-demand MBCT PD prevention intervention that is integrated within maternal clinical care settings using an existing patient portal. Successful achievement of the study aims will result in a refined implementation protocol for future studies that are sufficiently powered to evaluate the effectiveness of an integrated Digital Mental Health Technology and to estimate the cost/benefit ratio

DETAILED DESCRIPTION:
This type1 hybrid effectiveness-implementation project is conducted within healthcare settings and underserved populations (rural, urban, and Latino) and for individuals who are at risk for perinatal depression (PD), which allows the team to refine the approach in preparation for a future effectiveness trial for the prevention of PD in diverse communities using accessible Digital Mental Health Technology (patient education portal, FB discussion boards, synchronous videoconference support sessions). The plan is to adopt a randomized preference trial design to assess the impact of patient preference and sociocultural factors (including race, ethnicity, and geographic residence) on engagement and preliminary results. This information is crucial for a subsequent trial and for ultimately taking the intervention to scale. The study design using the IRLM reflects scientific rigor that can be reproduced by other investigators. The implemented strategies specifically developed to optimize implementation success, and to measure the implementation outcomes of these strategies and include valuable input from key informants, stakeholders, and the Community Advisory Board at regular intervals throughout the project time period.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age, who at the time of screening
* Have a viable pregnancy or are postpartum (up to 1 year)
* Identified as at-risk for PD (any one of the following:
* EPDS score equal to or greater than 9 or less than 21
* History of depression/anxiety
* 2 or more significant life events)
* English- or Spanish-speaking
* Currently attending a UHealth clinic or rural public health partner clinic.

Exclusion Criteria:

* Have a substance use disorder
* Current diagnosis of serious mental illness, such as psychosis, schizophrenia, bipolar disorder, severe depression (including EPDS > 20)
* Severe anxiety, suicidality, or currently taking any medications for a mental health condition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant and or postpartum women
Enrollment: 120 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Implementation outcome; Feasibility and acceptability | (6, 12 & 18 months)
  EPDS Scores are between 0 and 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder. Using scores that are between 9-20 Qualitative; semi structured interview Quantitative; patient satisfaction survey, number of referrals for at-risk patients, patients registering on YoMingo. focus groups, individual interviews, questionnaires

SECONDARY OUTCOMES:
Sociocultural Determinants and Behavior | 6, 12 & 18 months)
  EPDS Scores are between 0 and 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder.- using EPDS score between 9-20. Life events, cultural/ethnical/racial group membership, history of depression, mental stigma

OTHER OUTCOMES:
Implementation Outcome; Patient engagement | 6, 12 & 18 months)
  EPDS screening- Scores are between 0 and 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder. Using score 9-13. Evaluate preference & engagement in an 8-week remote-access MBCT or a program;;multimedia on- demand (OD) alone, or OD with a facilitated discussion board (DB) or OD with facilitated, synchronous videoconference sessions (VC).
Exploratory analysis of patient symptom | 6, 12 & 18 months)
  EPDS Scores are between 0 and 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder. Usinf score 9-20. Conduct an exploratory analysis of PD symptom trajectory for all paired study groups. The Edinburgh Postnatal Depression Scale (EPDS) will be completed at five timepoints (pre- and post- intervention, and 2-, 4-, and 6-months post-intervention) to model change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Latendresse, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

DOCUMENTS (1):
  • Informed Consent Form (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT06049433/ICF_000.pdf